CLINICAL TRIAL: NCT01902147
Title: Measuring Recovery in Patients Undergoing Major Abdominal, Thoracic, and Arthroplasty Surgery Using an Enhanced Recovery Program.
Brief Title: Postoperative Quality Recovery Scale (PQRS)
Status: Completed | Type: Observational
Sponsor: Franco Carli (Other)
Responsible Party: Sponsor-Investigator, Franco Carli, Professor, Department of Anesthesia, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Other Study IDs: 13-141-SDR
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Surgery; Recovery
Keywords: abdominal; thoracic; arthroplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elective major abdominal, thoracic, and arthroplasty surgery: All consenting patients scheduled for elective major abdominal, thoracic, and arthroplasty surgery will be followed for 8 weeks after surgery to measure the quality of recovering using the PQRS.
  Interventions: Other: Postoperative Quality Recovery Scale (PQRS)

INTERVENTIONS:
Other: Postoperative Quality Recovery Scale (PQRS) — The PQRS is completed prior to surgery to provide baseline values, and then repeated at different intervals: 15 minutes, 40 minutes, 1 and 3 days, and 4-8 weeks after the completion of surgery. Recovery is broadly defined as return to baseline or better.

SUMMARY:
Recovery following general anesthesia and surgery is a complex issue confounded by the type of surgery, surgical care, inflammation, different anesthetic drugs and techniques, patient co-morbidities, and differing patient and clinician perceptions of what constitutes good recovery. In this observational study, quality of recovery and patient satisfaction will be measured using the Postoperative Quality Recovery Scale (PQRS). This tool includes six domains of recovery: physiological, nociceptive (pain and nausea), emotive (anxiety and depression), functional recovery (return of activities of daily living), self-assessed recovery, and cognitive recovery.

ELIGIBILITY:
Inclusion Criteria:

* elective major abdominal, thoracic, and arthroplasty surgery

Exclusion Criteria:

* Poor comprehension of English or French

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing elective major abdominal, thoracic, and arthroplasty surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Incidence of recovery (return to baseline or better) in the cognitive domain of the PQRS | postoperative day 3

CONTACTS AND LOCATIONS:
Overall Officials: Franco Carli, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Royse CF, Newman S, Chung F, Stygall J, McKay RE, Boldt J, Servin FS, Hurtado I, Hannallah R, Yu B, Wilkinson DJ. Development and feasibility of a scale to assess postoperative recovery: the post-operative quality recovery scale. Anesthesiology. 2010 Oct;113(4):892-905. doi: 10.1097/ALN.0b013e3181d960a9. PMID 20601860